CLINICAL TRIAL: NCT04841031
Title: Psychosocial and Economic Impacts of Narrative Exposure Therapy for Violence Survivors in Eastern DRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: World Bank (Other)
Collaborators: Fonds Social de la République Démocratique du Congo (Unknown); Vivo international e.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P147489
Record Dates: First submitted 2020-05-07; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Mental Health Disorder; PTSD; Depression Anxiety Disorder; Gender-based Violence
MeSH Terms: conditions — Mental Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NET Treatment (Experimental): Narrative Exposure Therapy (NET) Treatment: Treatment group consists of eligible individuals who are randomly assigned to receive NET treatment and are part of the study sample. Within each health center, treated individuals are randomly selected over several cohorts. In every cohort, the treatment group contained 6 individuals who received NET.
  Interventions: Behavioral: NET Treatment
- Control (Other): This group contains eligible individuals who are randomly assigned to the control group and are part of the study sample. In every cohort, the control group contained 6 individuals.
  Interventions: Other: Alternative Intervention

INTERVENTIONS:
Behavioral: NET Treatment — Narrative Exposure Therapy (NET) aims to address PTSD symptoms among survivors of mass violence and torture (Onyut et al., 2004; Schauer, et al., 2005). Mainly, different from other psychosocial interventions which require the survivor to process a single traumatic event in his or her life at a given time, NET treatment recognizes that trauma survivors undergo multiple distressing events within their lifetime (Schauer et al., 2005). Focusing on the traumatic events, the patient constructs a chronological narrative of his or her life story and a coherent narrative is then structured with the assistance of the therapist. They received NET one to three months following their screening and randomization. The therapy involves 8 to 12 individual sessions of about 90 minutes each.
  Arms: NET Treatment
Other: Alternative Intervention — Individuals in control group received non-NET psychosocial support in the interim that is provided to SGBV survivors as part of the Great Lakes SGBV project and will then receive NET after endline data has been collected.
  Arms: Control

SUMMARY:
The objective of the study is to evaluate the impact of Narrative Exposure Therapy (NET) delivered by local counselors, on the mental health and socio-economic empowerment of survivors of Sexual and Gender Based Violence (SGBV) who suffer Post-Traumatic Stress Disorder (PTSD), in North and South Kivu in Eastern DRC. The counselors will be trained and supervised by clinical experts from the NGO Vivo International. The therapy is expected to reduce the symptoms of PTSD, depression, and anxiety in SGBV survivors. The project is expected to directly impact and improve the beneficiaries' mental health outcomes of interest, and to indirectly impact and enhance their economic empowerment in the medium term and social functioning both in the short and medium term. This proposed impact evaluation will answer the following research questions: 1) What is the impact of NET on survivors' psychosocial wellbeing, economic empowerment and social functioning and participation? 2) Does the impact of NET differ depending on individual and household characteristics as well as context-specific factors?

ELIGIBILITY:
Inclusion Criteria:

* GBV survivors who are screened for commonly found conditions of mental distress

Exclusion Criteria:

* More severe cases of mental disorders are ineligible. They are referred to the General Referral Hospitals or specialized mental health clinics to receive immediate treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1053 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2021-02-14 (Actual); Study Completion 2021-02-14 (Actual)

PRIMARY OUTCOMES:
Post-traumatic Stress Disorder (PTSD) Severity | Baseline, 3 months follow-up, 12 months follow-up
  Change in self-report experience of PTSD symptoms, assessed by using the Harvard Trauma Questionnaire (HTQ-16). This indicator will be constructed as the average PTSD severity score taking the average of the 16 items in HTQ-16 with a range from 0 to 3, where higher scores indicate worse symptoms.
Depression and Anxiety | Baseline, 3 months follow-up, 12 months follow-up
  Change in self-report experience of depression and anxiety symptoms, assessed by using the Hopkins Symptom Checklist-25 (HSCL-25). This indicator will be the average of 16 items, ranging from 0 to 3 where higher score indicates greater severity of depression or anxiety.

SECONDARY OUTCOMES:
Self-esteem | Baseline, 3 months follow-up, 12 months follow-up
  Change in self-reported measure of self-esteem, assessed using Rosenberg Self-Esteem Scale with 10 items that are rated on a 4-point Likert Scale (minimum value:0 and maximum value:3). After reversing the negative items, the self-esteem index will be constructed as the average of the per-item scores, higher scores indicating higher self-esteem.
Management of problems | Baseline, 3 months follow-up, 12 months follow-up
  Change in self-reported measure of management of problems in certain activities when they feel bad, such as talking to friends, family, other women with similar things, praying, working, locking herself in the house, drinking alcohol, singing, spending time with others. . After reversing the negative items, the index for management of problems will be constructed by taking the average of the values of the 8 items. The items are rated on a 4-point Likert Scale, with item values ranging from "0=Not at all/Never" to "3=Often". Higher scores will indicate improved management of problems (minimum value:0 and maximum value:3).
Local functioning impairment index | Baseline, 3 months follow-up, 12 months follow-up
  Change in self-reported experience of difficulties in performing certain activities, specifically to what extent they are experiencing difficulties in performing activities, such as farming, income generating activities, housework, socializing with family and community members, focusing on their tasks and responsibilities, cooking, taking care of children, exchange ideas, do any type of manual work, receive help, make important decisions, learn new skills, and interact with people they don't know in the last 4 weeks. The local functioning impairment index will be created by taking the average of 14 item scores rated on a 5-point Likert scale with values ranging from "0=No difficulty" to "4=So difficult that she couldn't do it". Higher scores will indicate greater impairment in local functioning (minimum value:0 and maximum value:4)
Labor force participation | Baseline, 3 months follow-up, 12 months follow-up
  Changes in the participation of respondents in income generating activities in the last 7 days. This indicator will be constructed as binary variable equal to 1 if the respondent reported any kind of work in the last 7 days, such as paid in-kind, unpaid, self-employment, non-farm family business or family farm.
Total Earnings | Baseline, 3 months follow-up, 12 months follow-up
  Change in the respondent's total earnings in the last 30 days (in main and secondary activities) in USD. This indicator will be the sum of the respondent's earnings from her main and secondary activities in the last 30 days.
Saving behavior | Baseline, 3 months follow-up, 12 months follow-up
  Changes in the number of participants who saved in the last 6 or 12 months.
Total amount of savings | Baseline, 3 months follow-up, 12 months follow-up
  Changes in the total amount of savings (formal or informal) in the last 6 or 12 months.
Decision-making power | Baseline, 3 months follow-up, 12 months follow-up
  Changes in the power of decision of the participant. We will create a power of decision index capturing the respondent's weight in making decisions regarding 1) her own income, 2) pregnancy, 3) children's education, 4) her own health care, 5) household money, 6) major purchases, and 7) visits to her family. We will construct the index by taking the mean of the items, where a higher score indicates more power of decision making. The range is [0-2].
Food insecurity | Baseline, 3 months follow-up, 12 months follow-up
  Changes in the number of average number of meals that the members of the respondent's household had to skip in the past 7 days, conditional on anyone in the household having to skip meal because there was not enough food.
Sharing of housework | Baseline, 3 months follow-up, 12 months follow-up
  Changes in the average score of the level of the participation of the respondent's partner in the domestic tasks. We will create this indicator as the average score of the level of the participation of the respondent's partner in the tasks of cooking and laundry-cleaning. First, we will score the partner's participation per task. Then we will create the index by taking the average score over the two tasks. The index will have a range of [0-3] with higher scores indicating more participation of the partner.
Respondent and household asset ownership | Baseline and 12 months follow-up
  Changes in the number of items owned by the respondent and the household

CONTACTS AND LOCATIONS:
Overall Officials: Julia Vaillant, PhD, Principal Investigator — World Bank
Locations (2):
- Democratic Republic of the Congo (2):
  - South Kivu, Bukavu
  - North Kivu, Goma

IPD SHARING:
Plan to Share IPD: Yes
The World Bank has an open data policy, and the de-identified, anonymized data will be published online after the study is completed.